CLINICAL TRIAL: NCT05579444
Title: Systems Biology of Gastrointestinal and Related Diseases
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment.
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Other Study IDs: V263
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Ulcerative Colitis; Crohn Disease; Obesity; Colon Polyp; Eosinophilic Esophagitis; GERD; Gastro Esophageal Reflux; Barrett Esophagus; Esophageal Cancer; Gastritis; Gastric Ulcer; Duodenal Ulcer; Intestinal Metaplasia; Gastric Cancer; Lymphocytic Colitis; Microscopic Colitis; Celiac Sprue; IBS; Irritable Bowel Syndrome; SIBO; NAFLD; Gallstone Disease
Keywords: gastrointestinal disease; gastric upset
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Obesity; Colonic Polyps; Eosinophilic Esophagitis; Gastroesophageal Reflux; Barrett Esophagus; Esophageal Neoplasms; Gastritis; Stomach Ulcer; Duodenal Ulcer; Stomach Neoplasms; Colitis, Lymphocytic; Colitis, Microscopic; Celiac Disease; Irritable Bowel Syndrome; Non-alcoholic Fatty Liver Disease; Cholelithiasis; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (17):
- Ulcerative Colitis: Participants with ulcerative colitis.
- Crohn's Disease: Participants with Crohn's disease.
- Obesity: Participants that are obese.
- Colon Polyps: Participants with colon polyps.
- Eosinophilic esophagitis: Participants with Eosinophilic esophagitis
- Gastroesophageal Reflux Disease (GERD): Participants with Gastroesophageal Reflux Disease (GERD).
- Gastritis: Participants with gastritis.
- Gastric ulcers: Participants with gastric ulcers.
- Duodenal ulcers: Participants with duodenal ulcers.
- Intestinal metaplasia: Participants with intestinal metaplasia (risk factor for esophageal cancer).
- Gastric Cancer: Participants with gastric cancer.
- Lymphocytic/Microscopic Colitis: Participants with Lymphocytic/Microscopic Colitis.
- Celiac Sprue: Participants with Celiac Sprue.
- Irritable Bowel Syndrome (IBS): Participants with IBS.
- Small intestinal bacterial overgrowth (SIBO): Participants with SIBO.
- Non-alcoholic Fatty Liver Disease (NAFLD): Participants with NAFLD.
- Gallstone disease: Participants with Gallstone disease.

SUMMARY:
This is a longitudinal observational study on patients with gastrointestinal and related disease. The study will be conducted for at least 10 years, following each participant over time, as they either go through relapses and remissions, or progression of their disease.

DETAILED DESCRIPTION:
This is a longitudinal, observational study whose main goal is to identify the human and microbial determinants of gastrointestinal diseases. Molecular and metadata will be collected from a large study population at multiple time points. Machine learning will be applied to all data, and models will be evaluated for development of novel diagnostic and therapeutic tools.

ELIGIBILITY:
Inclusion criteria

* Any patient 18 years old or older that schedules a visit to WAGI clinics or endoscopy center
* Able to use electronic communications
* Able to communicate in English
* Consent to participate in the study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years old or older who visit WAGI for the following reasons:
  * Colonoscopy
  * Screening
  * Surveillance
  * Diagnostic Esophagogastroduodenoscopy (EGD) Screening Surveillance Diagnostic Initial consultation: differential diagnosis (including suspected and definitive diagnosis), disease management plan, diagnostic plan (laboratories, imaging, medical therapy, non-medical therapy)
  * Follow-up visits: same as the initial visit
  * Biologic infusions (can collect disease activity levels at the time)
  * Diagnosis of any gastrointestinal disease
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Identification of human determinants of gastrointestinal diseases. | Up to 10 years
  Identification of biomarkers that indicate gastrointestinal diseases.
Identification of microbial determinants of gastrointestinal diseases. | Up to 10 years
  Identification of microbial species that indicate gastrointestinal disease.

SECONDARY OUTCOMES:
Prediction of efficacy of biologics in treating IBD. | Up to 10 years.
  Prediction of the efficacy of a biologic medication against IBD based on molecular data and metadata.
Development of a molecular test for C. difficile infection (CDI) | Up to 10 years.
  Development of a molecular test for C. difficile infection (CDI)
Quantify change in microbial species over time post colonoscopy | Up to 10 years.
  Quantification of changes observed in the microbiome post colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, Principal Investigator — Viome
Locations (1):
- Viome Life Sciences, Bothell, Washington, United States